CLINICAL TRIAL: NCT02223039
Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of Multiple Doses of AbGn-168H Administered by Intravenous Infusion to Patients With Moderate to Severe Chronic Plaque Psoriasis (Randomised, Double-blind, Placebo-controlled)
Brief Title: A Study of Multiple Doses of AbGn-168H by Intravenous Infusion in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbGenomics B.V Taiwan Branch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014.002.01
Record Dates: First submitted 2014-05-22; First posted 2014-08-22 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
Keywords: Psoriasis; Dermatology; Monoclonal antibody
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AbGn-168H Low Dose (Experimental): Subject to receive low dose of AbGn-168H intravenously
  Interventions: Biological: AbGn-168H
- AbGn-168H High Dose (Experimental): Subject to receive high dose of AbGn-168H intravenously
  Interventions: Biological: AbGn-168H
- Placebo (Placebo Comparator): Subject to receive placebo intravenously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AbGn-168H — AbGn-168H monoclonal antibody
  Arms: AbGn-168H High Dose; AbGn-168H Low Dose
Biological: Placebo — Placebo of AbGn-168H
  Arms: Placebo

SUMMARY:
This is a phase II, randomised, double-blind, placebo-controlled, multiple-dose, multi-center study of AbGn-168H in subjects with moderate to severe chronic plaque psoriasis. The objectives of this study is to investigate efficacy, safety, tolerability, and pharmacokinetics (PK) of multiple doses of AbGn-168H administered intravenously to patients with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 (inclusive), males or females
2. Body weight < 140 kg
3. Patients with stable moderate to severe plaque-type psoriasis, no significant changes within the past 6 months, involving ≥ 10% body surface area, with disease severity PASI ≥ 10 at screening visit and visit 2.
4. Psoriasis disease duration of at least 6 months prior to screening
5. Patients must be candidates for systemic psoriasis treatment or phototherapy
6. Patient must give informed consent and sign an approved consent form prior to any study procedures
7. Females of childbearing potential must have a negative pregnancy test result prior to enrollment and agree to use a highly effective method of birth control during the study. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year).

Exclusion Criteria:

1. Patients with primary guttatae, erythrodermic, or pustular psoriasis and patients with drug-induced psoriasis
2. Evidence of current or previous clinically significant disease, medical condition other than psoriasis, or finding of the medical examination (including vital signs and ECG), that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied. (Psoriatic arthritis is not considered an exclusion)
3. HIV infection or a known HIV-related Malignancy.
4. Chronic or acute hepatitis B and C, or carrier status. Patient with anti-HBc Ab and undetectable anti-HBs Ab should also be excluded.
5. Tuberculosis or a positive Tuberculin Skin Test (TST) for tuberculosis. Subjects previously received BCG vaccination or cannot receive TST can participate in the study after showing negative responses in Interferon-Gamma Release Assays (IGRA).
6. History of malignancy in the past 5 years or suspicion of active malignant disease except treated cutaneous squamous cell or basal cell carcinoma and carcinoma in situ of the cervix uteri.
7. History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
8. Use of biologic agents or investigational drug within 8-12 weeks prior to treatment, systemic anti-psoriatic medications or phototherapy within 4 weeks prior to treatment, or topical anti-psoriasis medications (except emollients) within 2 weeks prior to treatment
9. Intake of restricted medications or other drugs considered likely to interfere with the safe conduct of the study
10. Current alcohol abuse
11. Current drug abuse or positive drug screen at screening visit. Subjects with legitimate medically supervised uses of the drugs which are not excluded for other reasons can be enrolled.
12. Any blood donation or significant blood loss within 4 weeks prior to Visit 2
13. Excessive (e.g. competitive) physical activities (within 1 week prior to administration or during the trial)
14. Patients with any of the following laboratory values at screening and are considered clinically significant by the investigators:

    * Haemoglobin, hematocrit, white blood cell count, absolute lymphocyte or neutrophil count, or platelet count < LLN (below the lower limit of the reference normal range)
    * ALT, AST and/or total bilirubin > 2.5xULN
    * Serum creatinine > 1.5x ULN
15. Any clinically significant laboratory abnormalities other than those listed on Exclusion Criteria 14, based on the investigator's medical assessment at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
75% reduction in the Psoriasis Area Severity Index (PASI 75) | at week 10
  The primary objective of this study is to investigate efficacy of AbGn-168H in patients with moderate to severe chronic plaque psoriasis following intravenous administration of multiple doses compared to placebo.

SECONDARY OUTCOMES:
Number of participants with abnormal Physical Examination finding | At different time point for 20 weeks after the first treatment
Cmax | 12 weeks after the first treatment
  Individual Cmax and tmax values will be directly determined from the plasma concentration time profiles of each subject
Number of participants with Vital Sign change | At different time point for 20 weeks after the first treatment
Number of participants with abnormal ECG finding | At different time point for 20 weeks after the first treatment
Number of participants with abnormal Clinical Laboratory parameters | At different time point for 20 weeks after the first treatment
  blood chemistry, hematology and urinalysis
Number of participants with Adverse Event | At different time point for 20 weeks after the first treatment
T1/2 | At different time point for 12 weeks after the first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao Lin, MD, Ph.D, Study Director — AbGenmics B.V. Taiwan Branch; Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (15):
- United States (15):
  - Alliance Dermatology & MOHS Center, PC, Phoenix, Arizona
  - Northwest AR Clinical Trials Center, PLLC., Rogers, Arkansas
  - Renstar Medical Research, Ocala, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Progressive Medical Research, Tampa, Florida
  - DawesFretzin Clinical Research Group, LLC., Indianaopolis, Indiana
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - High Point Clinical Trials Cente, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Radiant Research, Inc., Greer, South Carolina
  - Suzanne Bruce and Associates, P.A., The Center for Skin Research, Katy, Texas
  - University of Utah Dermatology School of Medicine Dermatology 4A330, Salt Lake City, Utah